CLINICAL TRIAL: NCT00628264
Title: Safety, Tolerability and Pharmacodynamics of AP214 Acetate in Patients Undergoing Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to a considerably lower recruitment rate than anticipated
Sponsor: Action Pharma A/S (Industry)
Responsible Party: Action Pharma A/S, Action Pharma A/S
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AP214-CS004
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass Grafting; Valve Surgery; Kidney Injury
Keywords: cardiac surgery; coronary artery bypass grafting; valve surgery; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP214 (Experimental)
  Interventions: Drug: AP214
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP214 — Three AP214 bolus infusions administered over 10 minutes (prior to skin incision, at time of clamp-release and 6 hours after clamp-release).
  Arms: AP214
Drug: Placebo — Three placebo bolus infusions administered over 10 minutes (prior to skin incision, at time of clamp-release and 6 hours after clamp-release).
  Arms: Placebo

SUMMARY:
The purpose of the present research study is to investigate for the first time, the safety and tolerability of infusion doses of AP214 in subjects having heart surgery such as coronary bypass graft and/or valve repair or replacement surgery. AP214, the investigational drug, is being developed to potentially prevent post-surgical kidney injury after thoracic aortic aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the trial specific informed consent form.
2. Patients ≥ 18 years old, male or female, not of childbearing potential (postmenopausal or permanently sterilized e.g., tubal occlusion, hysterectomy, bilateral salpingectomy), regardless of ethnicity.
3. Patients undergoing CABG, valve(s), CABG/valve and/or aortic root or ascending aortic aneurysm repair surgery.
4. Cleveland Clinic Renal Score ≥ 2 (higher than average risk for AKI).
5. EF ≥ 30%, evaluated within 2 months prior to screening visit.

Exclusion Criteria:

1. Cardiac surgery to be performed "off pump" without cardiopulmonary bypass.
2. Circulatory arrest in connection with aortic root or ascending aortic aneurysm repair surgery.
3. Confirmed or suspected endocarditis.
4. Requiring a reoperation on one of the valves within 3 months following the original valve surgical procedure.
5. Receiving Aprotinin during the trial, from Screening to Day 90.
6. Having undergone cardiovascular catheterization ≤ 48 hours prior to scheduled surgery.
7. Active peptic ulcer disease and gastritis.
8. Hemoccult positive stools, hematological, bleeding, and coagulation disorders.
9. Receiving dopamine at renal doses (2-4 mcg/kg/min), from Screening to Day 90.
10. S-Creatinine greater than 2.1 mg/dl.
11. Known or suspected hypersensitivity to the investigational medicinal product.
12. Known or suspected hypersensitivity to ondansetron or other selective 5-hydroxytryptamine 3 (5-HT3) receptor antagonists.
13. Current participation in any other interventional clinical trial.
14. Previously dosed with AP214.
15. Use of investigational medicinal products within the previous 6 months.
16. Body weight above 140 kg.
17. History of any organ transplant.
18. Women who are of childbearing potential, pregnant or breast-feeding.
19. Current abuse of alcohol or substance, according to the investigator's medical judgment
20. Has a mental incapacity or language barriers precluding adequate understanding of trial procedures.
21. Is considered by the Investigator unsuitable to participate in the trial for any other reason for instance due to a significant serious underlying condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AP214 administered as three 10-minute bolus infusions, in patients undergoing cardiac surgery that are at increased risk of AKI (descriptive analysis of AEs and SAEs from Day 0-14). | From day 0-14
To assess the impact of AP214 on cardiac surgery induced systemic inflammatory response syndrome determined by the post-operative peak plasma concentrations of IL-6 and IL-10 from 0-24 hours | 0-24 hours

SECONDARY OUTCOMES:
To assess the safety and tolerability of AP214 at an organ level as well as in terms of the overall mortality (heart, CNS, lung, wound, mortality) | Day 0-90
To assess the impact of AP214 on cardiac surgery induced systemic inflammatory response syndrome (post-operative peak plasma concentrations of TNF-α and IL-8 and AUC for TNF-α, IL-6, IL-8 and IL-10). | 0-24 hours
To assess the impact of AP214 for renal protection as measured by the development of post-surgical acute kidney injury (AKIN score) | Day 0-14
To assess the impact of AP214 on the development of post-surgical left ventricular dysfunction (determined by changes in left ventricular function from pre to post coronary bypass by transesophageal echocardiography | 0-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Beaver, MD, MPH, Principal Investigator — Division of Thoracic and Cardiovascular Surgery , University of Florida College of Medicine
Locations (2):
- United States (2):
  - Shands Hospital at Alachua General Hospital, Gainesville, Florida
  - Shands Hopsital at University of Florida, Gainesville, Florida